CLINICAL TRIAL: NCT01132430
Title: Impact of a Motivational Interviewing Intervention on Medication Adherence in Patients With Asthma
Brief Title: Motivational Interviewing for Medication Adherence in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Simon Bacon, Co-PI, PI is Dr. Kim Lavoie, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBMC001
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2015-07

CONDITIONS: Asthma
Keywords: ADHERENCE; ASTHMA CONTROL; ASTHMA QUALITY OF LIFE; MOTIVATIONAL INTERVIEWING
MeSH Terms: conditions — Asthma | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Placebo Comparator): Standard medical care within 4-6 week period
  Interventions: Behavioral: Usual care
- Motivational interviewing (Experimental): Brief MI sessions within 4-6 week period
  Interventions: Behavioral: Motivational interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing — Brief MI 3x30 minute sessions within 4-6 week period
  Arms: Motivational interviewing
Behavioral: Usual care — Standard medical care within 4-6 week period
  Arms: Usual care

SUMMARY:
The high burden of asthma appears to be related to poor asthma control, which is associated with more frequent asthma symptoms, greater bronchodilator use and functional impairment, and worse pulmonary function. Despite the availability of effective treatments, more than 58% of asthmatics are poorly controlled. Daily adherence to inhaled corticosteroid (ICS) regimens is considered by experts to be one of the most important behavioral factors linked to achieving optimal asthma control. However, there is a paucity of research on interventions specifically designed to improve ICS adherence among adult asthmatics. The vast majority of intervention studies to date used atheoretical interventions to target behavior change, relying mainly upon educational approaches which have been criticised for "failing to translate knowledge into action." This may be due to the fact that most education-based approaches do not specifically address or help patients overcome ambivalence about behavior change, which is necessary for ensuring daily adherence. Motivational interviewing (MI) is a client-centred intervention that focuses on enhancing intrinsic motivation to change a particular behavior, and exploring and resolving ambivalence about behavior change. Brief MI sessions (e.g., 1-5 x 15-30 minute sessions) have been shown to improve a variety of health behaviors (e.g., reduce alcohol consumption, improve dietary habits, increase exercise behaviour, and improve medication adherence) and health outcomes (reduce blood pressure, body mass index, and cholesterol levels). However, no studies to date have assessed the efficacy of using MI to improve ICS adherence in asthmatics. This study aims to assess the efficacy of using MI to improve daily medication (ICS) adherence in a sample of poorly controlled, non-adherent asthmatics. It is hypothesized that patients randomized to the MI condition will exhibit significantly improved ICS adherence at 6 and 12-months post-intervention, independent of baseline levels and covariates, relative to patients randomized to the usual care control condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Primary diagnosis of moderate-severe persistent asthma (as per GINA)
* Prescribed inhaled corticosteroid medication (min dose of 250 µg fluticasone equivalent per day) for at least 12 consecutive months
* Uncontrolled asthma (≤ 19 on the Asthma Control Test)
* Covered by a drug insurance plan (e.g., RAMQ)
* Non-adherent to ICS medication (based on having filled less than 30% of their prescriptions over the last year)
* Able to speak English or French.

Exclusion Criteria:

* Any other medical condition that confers greater illness morbidity than asthma (e.g., active cancer)
* Severe psychopathology (e.g., schizophrenia)
* Apparent cognitive or language deficit
* Are or plan to become pregnant or move outside of Quebec over the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Inhaled corticosteroid adherence | 12 months post-intervention
  measured according to the following validated equation: # of treatment days (based on the # of canisters filled at the pharmacy x the duration of each prescription) divided by the # of prescription days (# of days the patient is expected to be taking his/her medication)

SECONDARY OUTCOMES:
Inhaled corticosteroid adherence | 6 months post-intervention
  measured according to the following validated equation: # of treatment days (based on the # of canisters filled at the pharmacy x the duration of each prescription) divided by the # of prescription days (# of days the patient is expected to be taking his/her medication)
Asthma Control Questionnaire (Juniper) | 12 months post-intervention, with preliminary data collected at 6 months
Asthma Control Test | 12 months post-intervention, with preliminary data collected at 6 months
Asthma Self-Efficacy Scale (Tobin) | 12 months post-intervention, with preliminary data collected at 6 months
Asthma Quality of Life Questionnaire (Juniper) | 12 months post-intervention, with preliminary data collected at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Lavoie, PhD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hopital du Sacre-Coeur de Montreal, Montreal, Quebec, Canada